CLINICAL TRIAL: NCT04608968
Title: Development and Validation of a Perioperative Satisfaction Questionnaire in Children Population
Brief Title: Pediatric Perioperative Satisfaction Questionnaire
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0346
Record Dates: First submitted 2020-09-24; First posted 2020-10-30 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Perioperative; Children; Satisfaction
Keywords: Validity; Questionnaire; Children; health quality of life; Self report
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to develop and validate a self-report questionnaire to evalutate the satisfaction of the children after surgery.

DETAILED DESCRIPTION:
Step 1 : development of the questiontionnaire Face to face interview to report the satisfaction of the children after surgery and to identify recurrent themes to generate questions.

Step 2 : validation of the questionnaire Evaluation of the psychometric validity of the final questionnaire

ELIGIBILITY:
Inclusion criteria:

* children 7 years and older
* elective surgery
* general anesthesia
* abiliy to understand and read questions

Exclusion criteria:

* emergency
* cognitive trouble
* intellectual disability

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children 7 years and older after surgery
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Children satisfaction after surgery | at discharge of hospital ( from the day of surgery up 14 days)
  to develop a questionnaire (score 0 to 100) to assess the satisfaction of children after surgery (from the day of surgery to 2 weeks)

SECONDARY OUTCOMES:
postoperative pain intensity | at discharge of hospital ( from the day of surgery up 14 days)
  to assess the level of children postoperative pain intensity (from the day of surgery to 2 weeks). Pain was assessed using the Face Pain Scale revised tool (0-10).
perioperative anxiety level | at discharge of hospital ( from the day of surgery up 14 days)
  to assess perioperative anxiety level using the Visual Analog Scale (0-10) of children after surgery (from the day of surgery to 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DADURE, PhD, Study Director — University Hospital, Montpellier
Locations (6):
- France (6):
  - Uhmontpellier, Montpellier, Montpellier
  - UH Bordeaux, Bordeaux
  - UH Grenoble, Grenoble
  - UH Nîmes, Nîmes
  - UH Reims, Reims
  - UH Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided
NC